CLINICAL TRIAL: NCT01759719
Title: Novara Platinum CROMium Everolimus EluTing StEnt SpontaneoUs RegiStry
Brief Title: Novara Registry of Platinum-Chromium Platform Stents
Acronym: PROMETEUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Lupi Alessandro, M.D., Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: 0000002
Record Dates: First submitted 2012-12-16; First posted 2013-01-03 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Fracture of Stent of Coronary Artery; External Causes of Morbidity and Mortality; Myocardial Infarction; Coronary Vessel Disorders
Keywords: platinum-chromium stents; concertina effect; stent deformation; everolimus eluting stents; stent lenght
MeSH Terms: conditions — Myocardial Infarction | interventions — Angioplasty, Balloon

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PtCr stent PCI treated patients: patients treated with PCI in whichat least 1 PtCr stent was used
  Interventions: Device: coronary angioplasty with PtCr stent implantation

INTERVENTIONS:
Device: coronary angioplasty with PtCr stent implantation — PCI with deployment of at least 1 PtCr stent
  Other Names: Promus Elements platinum Chromium stent; Omega platinum Chromium stent

SUMMARY:
Recent reports have described cases of novel thin-strut coronary stent longitudinal deformation during or after deployment and a biomechanical analysis have suggested increased susceptibility for such a complication for the platinum chromium (PtCr) coronary stent platforms . This analysis aims to assess the incidence of longitudinal stent deformation for PtCr stents in a large single centre all-comers population using quantitative angiographic analysis (QCA).

DETAILED DESCRIPTION:
Aims: Recent reports have described cases of novel thin-strut coronary stent longitudinal deformation during or after deployment and a biomechanical analysis have suggested increased susceptibility for such a complication for the platinum chromium (PtCr) coronary stent platforms .

The aim of this analysis is to assess the incidence of longitudinal stent deformation for PtCr stents in a large single centre all-comers population .

Methods: Quantitative angiographic analysis (QCA) of PtCr stents deployed in consecutive all-comers patients treated in our Laboratory from January 2011 to August 2012 will be performed by an independent core laboratory. In particular QCA : nominal stent lenght ratio will be calculated for every PtCr stent.

Clinical follow up with data about overall and cardiac mortality, myocardial infarction and target vessel revascularization will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* PCI with at least 1 platinum-chromium platform-based stent
* presence of at least 2 ortogonal angiographic projections of the deployed stent to allow proper quantitative coronary angiography

Exclusion Criteria:

* age <18 >90

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 253 consecutive all-comers patients treated in our Laboratory from January 2011 to August 2012 with PCI using a platinum-chromium platform based DES
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
QCA : nominal stent lenght ratio | 1 day
  QCA measured lenght of the deployed stent divided for the nominal stent lenght, a surrogate marker for stent deformation

SECONDARY OUTCOMES:
cardiovascular mortality | 1 year
  death from cardiac or vascular causes
myocardial infarction | 1 year
  recurring myocardial infarction (MI), according to the novel 3rd definition of MI
target vessel failure | 1 year
  any clinically-driver revascularization of the treated coronary vessel
Macroscopical stent deformation | 1 day
  severe stent deformation after deployment or other interventional manouvres (postdilation, IVUS, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Lupi, MD, Principal Investigator — AO Maggiore della Carita
Locations (1):
- Ospedale Maggiore della Carità, Novara, Piedmont, Italy

REFERENCES:
- [Derived] Lupi A, Porto I, Rognoni A, Lazzero M, Fattori R, Parisi R, De Maria GL, Bongo AS, Sheiban I, Bolognese L, Agostoni P, Secco GG; Novara-PROMETEUS (Platinum ChROMium Everolimus EluTing StEnt SpontaneoUs RegiStry) Investigators. Clinical and biomechanical behavior of a platinum-chromium stent platform in a large all-comer single-center population: insights from the Novara-PROMETEUS registry. J Invasive Cardiol. 2014 Jul;26(7):311-7. PMID 24993987